CLINICAL TRIAL: NCT01278940
Title: Phase I/II Trial of Vaccine Therapy With mRNA- Transfected Dendritic Cells in Patients With Advanced Malignant Melanoma
Brief Title: Trial of Vaccine Therapy With mRNA- Transfected Dendritic Cells in Patients With Advanced Malignant Melanoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Svein Dueland, MD, PhD, Oslo University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DC malignant melanoma
Record Dates: First submitted 2011-01-17; First posted 2011-01-19 (Estimated); Last update posted 2016-08-15 (Estimated); Status verified 2016-08

CONDITIONS: Malignant Melanoma
MeSH Terms: conditions — Melanoma | interventions — Interleukin-2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dendritic Cells (DC) malignant melanoma (Experimental): 22 patients were included in this arm.
  Interventions: Biological: Dendritic Cells (DC) malignant melanoma
- DC vaccine plus IL-2 (Experimental): To improve the efficacy of the DC vaccine, IL-2 was administrated at the vaccination site through direct lymph node injection. 9 patients were included in this arm.
  Interventions: Biological: Dendritic Cells (DC) malignant melanoma; Procedure: IL-2

INTERVENTIONS:
Biological: Dendritic Cells (DC) malignant melanoma — The patients were assigned to intradermal or intranodal DC vaccination
Procedure: IL-2 — IL-2 were administrated by intranodal injection
  Arms: DC vaccine plus IL-2

SUMMARY:
PRIMARY OBJECTIVES: Determination of safety and toxicity of vaccination with patients' tumour mRNA transfected DCs .

SECONDARY OBJECTIVES:Determine immunological response to the vaccine (induction of specific T-cell response) and assessment of tumour response

ELIGIBILITY:
Inclusion Criteria:

* Accessible tumour tissue for vaccine production (extraction of tumour mRNA) i.e.subcutaneous or lymph node metastases.
* Must be at least 18 years of age.
* Must have histologically confirmed advanced, metastatic cutaneous melanoma no longer amenable for surgery.
* Must have evidence of disease progression and measurable or evaluable metastases
* Must be ambulatory with a ECOG performance score of <2
* Must have lab.values as following :

ANC > 1.5 x 109/L; platelets > 100 x 109/L, Hb > 9g/dL (> 5.6 mmol/L). Creatinine < 140 µmol/L (1.6 mg/dL); if borderline, the creatinine clearance > 40 mL/min, Bilirubin < 20% above the upper limit of normal, ASAT and ALAT < 2.5 the upper limit of normal. Albumin > 2.5 g/L.

* Prior radiotherapy: A minimum of 4 weeks (8 weeks in case of extensive radiotherapy) must have elapsed between the end of the prior radiotherapy and entry into the protocol.
* Prior chemotherapy: A minimum 4 weeks must have elapsed between the end of the prior chemotherapy and entry into the protocol.
* Signed informed consent of the patients for the treatment and follow up must be obtained and documented according to the ICH-GCP Guidelines.

Exclusion Criteria:

* History of prior malignancy other than melanoma, with the exception of curatively treated basal cell or squamous cell carcinoma of the skin and ca. cervix stage 1B.
* Active infection requiring antibiotic therapy.
* Significant cardiac or other medical illness that would limit activity or survival, such as severe congestive heart failure, unstable angina, or serious cardiac arrhythmia.
* Autoimmune disease currently treated with steroids.
* Adverse reactions to vaccines such as anaphylaxis or other serious reactions.
* History of immunodeficiency or autoimmune disease such as rheumatoid arthritis, systemic lupus erythematosus, scleroderma, polymyositis-dermatomyositis, juvenile onset insulin dependent diabetes, or a vasculitic syndrome.
* Chemotherapy or other potentially immune-suppressive therapy that has been administered within 4 weeks prior to vaccination.
* Pregnancy or lactation.
* Any reason why, in the opinion of the investigator, the patient should not participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2002-03; Primary Completion 2006-02 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Determination of safety and toxicity of vaccination with patients' tumour mRNA transfected DCs | Patients are coming every week during 6 weeks.
  Biochemistry and hematology results, vital signs and ECOG performance status are measured at those timepoints.

SECONDARY OUTCOMES:
Determine immunological response to the vaccine (induction of specific T-cell response) | 6 weeks and 3 months after study start
Assessment of tumour response. | 3 months after study start
  CT-scan

CONTACTS AND LOCATIONS:
Overall Officials: Steinar Aamdal, M.D PhD Prof, Principal Investigator — Oslo University Hospital - Norwegian Radium Hospital

REFERENCES:
- [Result] Kyte JA, Mu L, Aamdal S, Kvalheim G, Dueland S, Hauser M, Gullestad HP, Ryder T, Lislerud K, Hammerstad H, Gaudernack G. Phase I/II trial of melanoma therapy with dendritic cells transfected with autologous tumor-mRNA. Cancer Gene Ther. 2006 Oct;13(10):905-18. doi: 10.1038/sj.cgt.7700961. Epub 2006 May 5. PMID 16710345
- [Result] Kyte JA, Kvalheim G, Lislerud K, thor Straten P, Dueland S, Aamdal S, Gaudernack G. T cell responses in melanoma patients after vaccination with tumor-mRNA transfected dendritic cells. Cancer Immunol Immunother. 2007 May;56(5):659-75. doi: 10.1007/s00262-006-0222-y. Epub 2006 Sep 1. PMID 16947019